CLINICAL TRIAL: NCT02231242
Title: Intrathecal Autologous Stem Cells for Children With Cerebral Palsy Phase II
Brief Title: Intrathecal Stem Cells for Cerebral Palsy Phase II
Acronym: ISCII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Consuelo Mancias Guerra, Dra. Consuelo Mancias Guerra, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: HE13-004
Record Dates: First submitted 2014-07-14; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Cerebral Palsy
Keywords: brain; children; cerebral palsy; bone marrow stem cells; intrathecal autologous total nucleated cells; quadriparesis
MeSH Terms: conditions — Cerebral Palsy; Quadriplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal Autologous Bone Marrow TNC (Experimental): Procedure/Surgery: Intrathecal Autologous Bone Marrow TNC. Other Names: Autologous Stem Cell Transplantation Patients will be stimulated with Granulocyte Colony Stimulating Factor (G-CSF) (10mcgr/kg of body weight) for 3 consecutive days. Bone marrow will be harvested under sedation and, after being processed in the laboratory, the autologous TNC concentrate of 10 mL will be infused intrathecally.
  Interventions: Biological: Autologous Stem Cell Transplantation
- Control group (No Intervention): Patients will be evaluated with the "Gross Motor Functional Classification System" initially, at one, three and six months, and then cross to the intervention arm.

INTERVENTIONS:
Biological: Autologous Stem Cell Transplantation — Patients will be stimulated with Granulocyte Colony Stimulating Factor (G-CSF) 3 consecutive days. Bone marrow will be harvested under sedation and, after being processed in the laboratory, the buffy coat (TNC) of 10 mL will be infused intrathecally.
  Intrathecal Autologous Bone Marrow TNC
  Arms: Intrathecal Autologous Bone Marrow TNC

SUMMARY:
The purpose of this study is to determine whether the infusion of intrathecal autologous bone marrow total nucleated cells would improve the neurologic evolution of pediatric patients with quadriparetic cerebral palsy.

DETAILED DESCRIPTION:
There is accumulated evidence that shows that the administration of bone marrow total nucleated cells (TNC) into the brain may produce some benefits by different mechanisms like cytokine production, in several neurological areas such as motor, social, adaptative and cognitive.

It has been found that after introducing TNC in the subarachnoid space of the spinal cord, these cells may be transported through the cerebrospinal fluid and can be delivered more efficiently to the injured area, compared with intravenous route in patients with neurologic injury.

Patients will be stimulated for 3 consecutive days with subcutaneous granulocyte colony stimulating factor (G-CSF) and then their bone marrow will be harvested according to their weight. Bone marrow will be processed in order to obtain the buffy coat and minimize the amount of red blood cells. An inoculum of 10mL of this TNC will be infused intrathecally. Patients will be evaluated with the "Gross Motor Functional Classification System" before the procedure and one, three and six months after that.

ELIGIBILITY:
Inclusion Criteria:

* Patients with quadriplegic cerebral palsy, with an age from 7 to 9 years of age, regardless the age at the time of injury, time post-injury, or previously received therapies, different from ours

Exclusion Criteria:

* Patients with neurodegenerative or autoimmune diseases
* Patients with active infection in any organ or tissue at the time of entering the study, the onset of stimulation with G-CSF or at the procedure
* Patients who do not sign the informed consent form

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants who show progress in GMFCS scale after autologous bonemarrow TNC intrathecal infusion. | six months
  Patients, in an outpatient basis, will be stimulated with Granulocyte Colony Stimulating Factor (G-CSF) for 3 consecutive days. Their bone marrow will be harvested under sedation and, after being processed in the laboratory, the buffy coat of 10 mL will be infused intrathecally.
  Patient will be monitored during acute phase to register any adverse effect (malaise, headache, fever, and nausea or vomit, etc).Gross Motor Function Classification System (GMFCS) scale is going to be monitored at baseline, one, three and six months to measured differences between the scales.
  GMFCS is based on patient's self-initiated movement with particular emphasis on sitting, walking, and wheeled mobility. Distinctions between levels are based on functional abilities, the need for assistive technology, including hand-held mobility devices (walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo Mancias-Guerra, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Hematology Service, Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Mancias-Guerra C, Marroquin-Escamilla AR, Gonzalez-Llano O, Villarreal-Martinez L, Jaime-Perez JC, Garcia-Rodriguez F, Valdes-Burnes SL, Rodriguez-Romo LN, Barrera-Morales DC, Sanchez-Hernandez JJ, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Gomez-De Leon A, Elizondo-Riojas G, Salazar-Riojas R, Gomez-Almaguer D. Safety and tolerability of intrathecal delivery of autologous bone marrow nucleated cells in children with cerebral palsy: an open-label phase I trial. Cytotherapy. 2014 Jun;16(6):810-20. doi: 10.1016/j.jcyt.2014.01.008. Epub 2014 Mar 15. PMID 24642016
- [Background] Mehta T, Feroz A, Thakkar U, Vanikar A, Shah V, Trivedi H. Subarachnoid placement of stem cells in neurological disorders. Transplant Proc. 2008 May;40(4):1145-7. doi: 10.1016/j.transproceed.2008.03.026. PMID 18555135
- [Background] Pakula AT, Van Naarden Braun K, Yeargin-Allsopp M. Cerebral palsy: classification and epidemiology. Phys Med Rehabil Clin N Am. 2009 Aug;20(3):425-52. doi: 10.1016/j.pmr.2009.06.001. PMID 19643346
- [Background] Felling RJ, Snyder MJ, Romanko MJ, Rothstein RP, Ziegler AN, Yang Z, Givogri MI, Bongarzone ER, Levison SW. Neural stem/progenitor cells participate in the regenerative response to perinatal hypoxia/ischemia. J Neurosci. 2006 Apr 19;26(16):4359-69. doi: 10.1523/JNEUROSCI.1898-05.2006. PMID 16624956
- [Background] Eglitis MA, Mezey E. Hematopoietic cells differentiate into both microglia and macroglia in the brains of adult mice. Proc Natl Acad Sci U S A. 1997 Apr 15;94(8):4080-5. doi: 10.1073/pnas.94.8.4080. PMID 9108108
- [Background] Woodbury D, Schwarz EJ, Prockop DJ, Black IB. Adult rat and human bone marrow stromal cells differentiate into neurons. J Neurosci Res. 2000 Aug 15;61(4):364-70. doi: 10.1002/1097-4547(20000815)61:43.0.CO;2-C. PMID 10931522
- [Background] Mezey E, Key S, Vogelsang G, Szalayova I, Lange GD, Crain B. Transplanted bone marrow generates new neurons in human brains. Proc Natl Acad Sci U S A. 2003 Feb 4;100(3):1364-9. doi: 10.1073/pnas.0336479100. Epub 2003 Jan 21. PMID 12538864
- [Background] Hayashi T, Iwai M, Ikeda T, Jin G, Deguchi K, Nagotani S, Zhang H, Sehara Y, Nagano I, Shoji M, Ikenoue T, Abe K. Neural precursor cells division and migration in neonatal rat brain after ischemic/hypoxic injury. Brain Res. 2005 Mar 15;1038(1):41-9. doi: 10.1016/j.brainres.2004.12.048. PMID 15748871
- [Background] Nakatomi H, Kuriu T, Okabe S, Yamamoto S, Hatano O, Kawahara N, Tamura A, Kirino T, Nakafuku M. Regeneration of hippocampal pyramidal neurons after ischemic brain injury by recruitment of endogenous neural progenitors. Cell. 2002 Aug 23;110(4):429-41. doi: 10.1016/s0092-8674(02)00862-0. PMID 12202033
- [Background] Rempe DA, Kent TA. Using bone marrow stromal cells for treatment of stroke. Neurology. 2002 Aug 27;59(4):486-7. doi: 10.1212/wnl.59.4.486. No abstract available. PMID 12196638
- [Background] Li Y, Chen J, Chen XG, Wang L, Gautam SC, Xu YX, Katakowski M, Zhang LJ, Lu M, Janakiraman N, Chopp M. Human marrow stromal cell therapy for stroke in rat: neurotrophins and functional recovery. Neurology. 2002 Aug 27;59(4):514-23. doi: 10.1212/wnl.59.4.514. PMID 12196642
- [Background] Gordon PH, Yu Q, Qualls C, Winfield H, Dillon S, Greene PE, Fahn S, Breeze RE, Freed CR, Pullman SL. Reaction time and movement time after embryonic cell implantation in Parkinson disease. Arch Neurol. 2004 Jun;61(6):858-61. doi: 10.1001/archneur.61.6.858. PMID 15210522
- [Background] Kulbatski I, Mothe AJ, Nomura H, Tator CH. Endogenous and exogenous CNS derived stem/progenitor cell approaches for neurotrauma. Curr Drug Targets. 2005 Feb;6(1):111-26. doi: 10.2174/1389450053345037. PMID 15720218
- [Background] Back SA, Rivkees SA. Emerging concepts in periventricular white matter injury. Semin Perinatol. 2004 Dec;28(6):405-14. doi: 10.1053/j.semperi.2004.10.010. PMID 15693397
- [Background] Follett PL, Deng W, Dai W, Talos DM, Massillon LJ, Rosenberg PA, Volpe JJ, Jensen FE. Glutamate receptor-mediated oligodendrocyte toxicity in periventricular leukomalacia: a protective role for topiramate. J Neurosci. 2004 May 5;24(18):4412-20. doi: 10.1523/JNEUROSCI.0477-04.2004. PMID 15128855
- [Background] Levison SW, Rothstein RP, Romanko MJ, Snyder MJ, Meyers RL, Vannucci SJ. Hypoxia/ischemia depletes the rat perinatal subventricular zone of oligodendrocyte progenitors and neural stem cells. Dev Neurosci. 2001;23(3):234-47. doi: 10.1159/000046149. PMID 11598326
- [Background] Robinson S, Petelenz K, Li Q, Cohen ML, Dechant A, Tabrizi N, Bucek M, Lust D, Miller RH. Developmental changes induced by graded prenatal systemic hypoxic-ischemic insults in rats. Neurobiol Dis. 2005 Apr;18(3):568-81. doi: 10.1016/j.nbd.2004.10.024. PMID 15755683
- [Background] Goldman SA, Schanz S, Windrem MS. Stem cell-based strategies for treating pediatric disorders of myelin. Hum Mol Genet. 2008 Apr 15;17(R1):R76-83. doi: 10.1093/hmg/ddn052. PMID 18632701
- [Background] Herzog EL, Chai L, Krause DS. Plasticity of marrow-derived stem cells. Blood. 2003 Nov 15;102(10):3483-93. doi: 10.1182/blood-2003-05-1664. Epub 2003 Jul 31. PMID 12893756
- [Background] Goodell MA. Stem-cell "plasticity": befuddled by the muddle. Curr Opin Hematol. 2003 May;10(3):208-13. doi: 10.1097/00062752-200305000-00003. PMID 12690288
- [Background] Appel SH, Engelhardt JI, Henkel JS, Siklos L, Beers DR, Yen AA, Simpson EP, Luo Y, Carrum G, Heslop HE, Brenner MK, Popat U. Hematopoietic stem cell transplantation in patients with sporadic amyotrophic lateral sclerosis. Neurology. 2008 Oct 21;71(17):1326-34. doi: 10.1212/01.wnl.0000327668.43541.22. PMID 18936424
- See also: web page — http://www.hematologia-uanl.com/